CLINICAL TRIAL: NCT05716919
Title: A Phase I, Double Blind, Randomized, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Orally Administered 'Ivaltinostat' Capsule in Healthy Male Volunteers
Brief Title: Multiple Ascending Dose Study of CG200745 'Ivaltinostat' Oral Capsule
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Machaon Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CG200745-1-02
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hematologic Malignancy; Solid Tumor; Fibrosis
MeSH Terms: conditions — Hematologic Neoplasms; Fibrosis | interventions — N1-(3-(dimethylamino)propyl)-N8-hydroxy-2-((naphthalene-1-loxy)methyl)oct-2-enediamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - 4 (Experimental): Cohort 1 : 50 mg/day Cohort 2 : 100 mg/day Cohort 3: 200mg/day [Cohort 4: 300mg/day: based on the result of Safety Review Meeting (SRM)]
  Interventions: Drug: Ivaltinostat
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivaltinostat — Ivaltinostat capsule
  Arms: Cohort 1 - 4
Other: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
A Phase I, Double blind, Randomized, Placebo-controlled, Multiple Ascending Dose Study to evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Orally Administered 'CG-745' Capsule in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria

1. Patients who are between 19 to 50 years of age at screening visit.
2. Patients who have body weight between 50.0 to 90.0 kg, and Body Mass Index (BMI) of 18.0 to 30.0 kg/m2 at screening visit.

   ☞ BMI (kg/m2) = Body Weight (kg) / {Height(m)}2
3. Patients who have signed informed consent prior to study participation after receiving detailed information on the purpose and details of the study, the characteristics of the test drug, and the expected adverse events.
4. Patients who are determined to be eligible by the investigator after evaluation of the following screening results: study questionnaires, physical examination, laboratory test, electrocardiogram, vital signs).

Exclusion Criteria

1. Medical history of clinically significant hepatic, renal, neurological, respiratory, endocrine, hematological, oncological, cardiovascular, urinary, and/or psychiatric disorder.
2. History of gastrointestinal disease or gastrointestinal surgery (except for simple appendectomy or hernia operation) that may affect the pharmacokinetic and/or safety evaluation of IP medications.
3. Known clinically significant hypersensitivity to HDAC inhibitors and/or other drugs.
4. Systolic blood pressure (SBP) less than 90 mmHg or over 140 mmHg; diastolic blood pressure (DBP) less than 50 mmHg or over 95 mmHg; pulse rate less than 45/min or over 100/min in the sitting position after a 5-minute rest.
5. Patients who show one or more of the following findings during screening (including additional tests):

   * AST (GOT) or ALT (GPT) exceeds 1.5 times the upper limit of the normal range ② Total bilirubin exceeds 1.5 times the upper limit of the normal range ③ Absolute neutrophil count (ANC) lower than 2,000/uL ④ Hb less than 12.5 g/dL ⑤ Platelets count less than 130,000/uL
6. Participation in another clinical study or bioequivalence study within 180 days prior to the first IP administration.
7. Positive result in serum tests (hepatitis B, hepatitis C, human immunodeficiency virus, and syphilis).
8. Donation of whole blood within 60 days, apheresis within 30 days, or transfusion within 30 days prior to the first IP administration.
9. Exposure to prescribed medications or herbal medicines 2 weeks prior to the first IP administration, or any general medication (OTC drug), health supplements, and/or vitamin supplements within 1 week prior to the first investigational product administration (the subject may still participate if the principal investigator determines that the subject is eligible for enrollment).
10. History of heavy smoking (more than 10 cigarettes/day) within three months prior to the first IP administration, or positive test result in urine cotinine test.
11. Excessive caffeine intake (> 5 units/day, 1 unit = 100 mg), excessive alcohol intake (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to abstain from drinking during admission period.
12. Inability to use a medically acceptable contraceptive method* for the duration of the study and up to 3 months after the last IP administration.

    * Medically acceptable contraception:
    * Use of intrauterine device (by spouse or partner) with a proven pregnancy prevention rate.
    * Concomitant use of barrier method (male or female) and spermicide.
    * Patient's or partner's surgery (vasectomy, salpingectomy, tubal ligation, or hysterectomy).
13. Patients who are determined to be ineligible to participate in the study by the principal investigator due to other reasons.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Plasma Pharmacokinetic measures (Cmax, Cmax-ss) | up to 4 weeks
Plasma Pharmacokinetic measures (AUC max, AUCmax-ss) | up to 4 weeks

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Serious or Non-Serious Adverse Events | Up to 4 weeks for each dosing cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea